CLINICAL TRIAL: NCT04251611
Title: Randomized Clinical Trial by Conglomerates on the Efficacy of the Maintenance of Physical Exercise for Patients With Myocardial Ischemia. Study Cardiopathy Prevention and Exercise in Phase 3 (CarPE3)
Brief Title: Randomized Clinical Trial by Conglomerates on the Efficacy of Maintenance of Physical Exercise in Myocardial Ischemia
Acronym: CarPE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Núria Santaularia Capdevila (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor-Investigator, Núria Santaularia Capdevila, Principal Investigator, Althaia Xarxa Assistencial Universitària de Manresa
Organization: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEIC 18/82
Record Dates: First submitted 2019-07-19; First posted 2020-02-05 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-06

CONDITIONS: Myocardial Ischemia; Physical Exercise
Keywords: Cardiac Rehabilitation; Myocardial Ischemia; Physical Exercise; Cardiovascular Risk Factors; Randomized Controlled Trial
MeSH Terms: conditions — Myocardial Ischemia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The usual care in patients with myocardial ischemia without other cardiovascular risk factors (CVFR) will be to attend one visit per year with doctor and nurse of the local health center. In this visit, it will be done a blood test and an electrocardiogram. Blood pressure, weight, body mass index, abdominal circumference will be measured and, in case of detecting enolic habit, smoking or sedentary lifestyle, generic advice will be done. If the patient, apart from myocardial ischemia, presents diabetes mellitus type 2, 3-4 follow-up visits per year will be recommended and will be increased according to specific needs. In case of presenting hypertension, will be recommended 2 visits with the nurse and one visit with the doctor per year and will be increased according to specific needs. In addition, in this case the blood pressure is checked every 6 months. During all visits, professionals will reinforce the control of CVRF and the maintenance of a long-term cardio-healthy lifestyle.
- Intervention group (Experimental): Patient will go to health center to visit the cardiac rehabilitation (CR) reference team, which is composed for a doctor and a nurse. This team will establish the guideline of action in the maintenance and/or increase in the physical exercise practice, in function of the resources of each zone and the preferences and motivations of the patient. They also reinforce the control of CVRF and the maintenance of a long-term cardio-healthy lifestyle.
  At the end of the visit, control visit will be given with the CR reference team at 3, 6 and 12 months after completing the supervised physical exercise program of phase II of the CRP. In case of detecting specific needs for the patient and/or relapses, the team will consult with the appropriate professional (cardiologist, cardiology nurse, physiotherapist, rehabilitator, nutritionist and/or psychologist). At the same time, the patient will be informed of the possibility of re-evaluating the CR reference team.
  Interventions: Other: Maintenance of physical exercise

INTERVENTIONS:
Other: Maintenance of physical exercise — Objectives will be established with the patient to increase the practice of physical exercise and reinforce the control of cardiovascular risk factors (CVRF) and the maintenance of a long-term cardio-healthy lifestyle.
  Other Names: Strengthen the control of cardiovascular risk factors
  Arms: Intervention group

SUMMARY:
Main objective: To assess the efficacy of a phase III cardiac rehabilitation program (CRP), based on counseling in the maintenance of physical exercise (time of physical exercise per week) for patients with myocardial ischemia (MI), once the supervised physical exercise program of phase II of CRP is completed.

Secondary objectives: To assess the efficacy of a phase III program of CRP based on counseling in the maintenance of physical exercise for the patient with MI in: 1) the energy expenditure per week, 2) body mass index and abdominal perimeter, 3) control of cardiovascular risk factors (smoking, high blood pressure, dyslipidemia and diabetes mellitus), 4) quality of life related to health, 5) assess the adherence to cardiac pharmacological treatment.

Method: Randomized clinical trial in conglomerates, open and controlled. The intervention group will carry out phase III of CRP based on counseling in the maintenance of physical exercise. The control group will receive the usual care. The main outcome will be the physical exercise time per week after finish the supervised physical exercise program of phase II of CRP and at 6 and 12 month later according to the 7-day Physical Activity Recall.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with myocardial ischemia, angina pectoris, other specific forms of chronic ischemic heart disease or unspecified ischemic heart disease.
* Patients who have completed the supervised physical exercise program of phase II of the CRP.
* Absence of cognitive deficit (Pfeiffer test: 0-2 mistakes).
* Sufficient functional capacity to follow the CRP (Barthel index >60)
* Residence in catchment area of Bages and Moianès.
* Providing signed informed consent.

Exclusion Criteria:

* Symptoms of right heart failure producing pulmonary hypertension.
* Dyspnea caused by severe pulmonary pathology.
* Additional comorbidities affecting the prognosis of cardiac disease.
* Major comorbidities or limitations that could interfere with the exercise training programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
The physical exercise minutes performed by the patient per week | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  The physical exercise minutes performed by the patient per week will be recorded through the 7-day Physical Activity Recall (PAR) questionnaire.
The physical exercise minutes performed by the patient per week | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  The physical exercise minutes performed by the patient per week will be recorded through the 7-day Physical Activity Recall (PAR) questionnaire.
The physical exercise minutes performed by the patient per week | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  The physical exercise minutes performed by the patient per week will be recorded through the 7-day Physical Activity Recall (PAR) questionnaire.

SECONDARY OUTCOMES:
The energy expenditure by the patient per week | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  The energy expenditure by the patient per week will be recorded through the 7-day Physical Activity Recall (PAR) questionnaire.
The energy expenditure by the patient per week | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  The energy expenditure by the patient per week will be recorded through the 7-day Physical Activity Recall (PAR) questionnaire.
The energy expenditure by the patient per week | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  The energy expenditure by the patient per week will be recorded through the 7-day Physical Activity Recall (PAR) questionnaire.
The body mass index (BMI) | At baseline of the supervised physical exercise program of phase II of the CRP has been completed.
  BMI is the quotient between the weight (kg) and the square of the height (m). It is usually used for the definition of underweight (BMI <15.99), normal weight (BMI 18.5 to 24.99), overweight (BMI ≥ 25 kg / m2) and obesity (BMI ≥ 30 kg / m2).
The body mass index (BMI) | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  BMI is the quotient between the weight (kg) and the square of the height (m). It is usually used for the definition of underweight (BMI <15.99), normal weight (BMI 18.5 to 24.99), overweight (BMI ≥ 25 kg / m2) and obesity (BMI ≥ 30 kg / m2).
The abdominal circumference | At baseline of the supervised physical exercise program of phase II of the CRP has been completed.
  Abdominal circumference is the measurement of the abdomen of the patient at the level of the navel. It will be recorded in centimeters using a tape measure.
The abdominal circumference | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Abdominal circumference is the measurement of the abdomen of the patient at the level of the navel. It will be recorded in centimeters using a tape measure.
The control of smoking | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Smoking:The degree of dependence on tobacco consumption will be recorded through the Fargeström test.
The control of smoking | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Smoking:The degree of dependence on tobacco consumption will be recorded through the Fargeström test.
The control of smoking | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Smoking:The degree of dependence on tobacco consumption will be recorded through the Fargeström test.
Systolic blood pressure | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Systolic blood pressure | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Systolic blood pressure | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Diastolic blood pressure | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Diastolic blood pressure | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Diastolic blood pressure | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Total cholesterol | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Total cholesterol | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Total cholesterol | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Low-density lipoproteins cholesterol | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Low-density lipoproteins cholesterol | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Low-density lipoproteins cholesterol | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
High-density lipoproteins cholesterol | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
High-density lipoproteins cholesterol | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
High-density lipoproteins cholesterol | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Triglycerides | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Triglycerides | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Triglycerides | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Basal plasma glucose | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Basal plasma glucose | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
Basal plasma glucose | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Physiological parameter
The quality of life related to health. | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  Level of perception of the patient regarding their state of health. It will be measured through the EuroQol-5D test.
The quality of life related to health. | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Level of perception of the patient regarding their state of health. It will be measured through the EuroQol-5D test.
The quality of life related to health. | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  Level of perception of the patient regarding their state of health. It will be measured through the EuroQol-5D test.
Assess the adherence to cardiovascular medication. | At baseline, when the supervised physical exercise program of phase II of the CRP has been completed.
  It will be recorded if the patient is successfully taking the cardiovascular medication through the Haynes-Sackett test.
Assess the adherence to cardiovascular medication. | At 6 months of the supervised physical exercise program of phase II of the CRP has been completed.
  It will be recorded if the patient is successfully taking the cardiovascular medication through the Haynes-Sackett test.
Assess the adherence to cardiovascular medication. | At 12 months of the supervised physical exercise program of phase II of the CRP has been completed.
  It will be recorded if the patient is successfully taking the cardiovascular medication through the Haynes-Sackett test.

CONTACTS AND LOCATIONS:
Overall Officials: Núria Santaularia, MSc, PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa
Locations (1):
- Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with a request of researchers. All the information will be anonymous.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When final results of the study will be published.
Access Criteria: Data will be shared with researchers or research team with a protocol study approved and/or with a clinical trial registred at a clinical trial register.